CLINICAL TRIAL: NCT04581889
Title: Prospective, Seroepidemiological, Non-invasive Cohort Study in Tübingen Children Age-stratified by Nursery and School Attendance
Brief Title: Prevalence of Antibodies Against SARS-CoV-2 Virus That Causes COVID-19 in Tübingen Children
Acronym: Coro-Buddy
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: Coro-Buddy
Record Dates: First submitted 2020-10-07; First posted 2020-10-09 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2022-06

CONDITIONS: Severe Acute Respiratory Syndrome
Keywords: SARS-CoV-2; antibodies; saliva; children; epidemiology
MeSH Terms: conditions — Severe Acute Respiratory Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Saliva, whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Children: Children from1 to 18 years, enrolled in kindergartens, primary, or secondary school located in city of Tübingen, Germany.
  Interventions: Other: Diagnostic test
- Adult comparator: Adults of unknown status of previous SARSCoV-2 infection.
- Adult validation: Adults who report a history of SARS-CoV-2 infections between 1. February 2020 and the time point of sampling.

INTERVENTIONS:
Other: Diagnostic test — Presence of antibodies in saliva
  Groups: Children

SUMMARY:
This is a prospective, longitudinal study to determine the incidence of SARS-COV-2 infection in children and adolescents by measuring specific antibodies in non-invasive saliva sampled in kindergartens and schools in a defined city area. The study includes an additional arm to validate the ELISA for anti-SARS-COV-2 reactive antibody measurements in saliva compared against blood collected in adult volunteers in a bimonthly follow-up period for 12 months.

DETAILED DESCRIPTION:
The world is confronting Coronavirus Disease-2019 (COVID-19) pandemic caused by SARS-CoV-2 virus, which is causing many deaths and burden on intensive care facilities. Data regarding epidemiologic characteristics in children and young adults is limited, especially in the context of educational settings. Due to mild symptoms or even asymptomatic cases in children, the rate of SARS-CoV-2 infected children is underestimated. Therefore, the present study aims to determine the incidence of SARS-CoV-2 infection in children at 3 timepoints during 12 months expressed as seroconversion measured in non-invasive saliva sampling in Tübingen, a defined study area. Children and adolescents (N = 1850) in the age of 1 to 17 years will be recruited via child-care, kindergarten and primary and secondary schools and followed-up for 12 months: shortly after release of lock-down measures in summer 2020, before winter and after the winter. An adult cohort (adult comparator group) is sampled at the same time points for incidence comparisons. To validate the ELISA for SARS-CoV-2 antibody measurements in saliva compared to blood, and to understand the half-life of SARS-CoV-2 antibodies in respective body fluids, peripheral blood and in saliva will be sampled every 2 months in an additional adult group (adult validation group).

ELIGIBILITY:
Inclusion Criteria:

* Children from 1 months to 18 years
* Written informed consent of the parent/legal guardian (study population is minor)
* Written assent when children are ≥ 12 years
* Enrolled in a kita, kindergarden, primary, or secondary school located in Tübingen

Adult population:

* Individuals >18 years who recovered from a confirmed SARS-CoV-2 infection.
* Or individuals > 18 years with an unknown status of previous SARS-CoV-2 infection

Exclusion Criteria:

* Unwilling to give consent

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Group A: Kita cohort (any age, usually 1-3 years): N = 350 Group B: Kindergarten cohort (any age, usually 3-6 years): N = 350 Group C: Primary school cohort (any age, usually, 6-10 years): N = 350 Group D: Secondary school, young cohort (class 5-8, any age, usually 10 - 14 years): N =400 Group E: Secondary school, adolescent cohort (class 9-12, any age, usually 14 - 18 years): N = 400 Group F: Tübinger adults (> 18 years): N = 400 (adult comparator group)
  Adults (n = 80). Specifically, 40 adult individuals who had a previous confirmed SARS-CoV-2 infection as well as 40 adults without previous SARS-CoV-2 infection at the start of the study.
Sampling Method: Probability Sample
Enrollment: 2380 (Actual)
Dates: Start 2020-07-02 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Incidence of SARS-CoV-2 infection in infants, children and adolescents | 12 months
  Identification of children that have been infected over different periods of time (summer, before winter and after winter) based on saliva samples

SECONDARY OUTCOMES:
Incidence of SARS-CoV-2 | 12 months
  Change of incidence of SARS-CoV-2 infection in children during 2020/2021

OTHER OUTCOMES:
SARS-CoV-2 antibody persistence | 12 months
  SARS-CoV-2 antibodies persistence in peripheral blood and saliva
Antibodies presence in saliva samples | 18 months
  Saliva samples as alternative for the detection of antibodies against SARS-CoV-2

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Kreidenweiss, Dr., Principal Investigator — University Hospital Tübingen; Jana Held, Dr, Principal Investigator — University Hospital Tübingen
Locations (1):
- Institute of Tropical Medicine, Tübingen, Deutschland, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hong H, Wang Y, Chung HT, Chen CJ. Clinical characteristics of novel coronavirus disease 2019 (COVID-19) in newborns, infants and children. Pediatr Neonatol. 2020 Apr;61(2):131-132. doi: 10.1016/j.pedneo.2020.03.001. Epub 2020 Mar 10. No abstract available. PMID 32199864
- [Background] Zimmermann P, Curtis N. COVID-19 in Children, Pregnancy and Neonates: A Review of Epidemiologic and Clinical Features. Pediatr Infect Dis J. 2020 Jun;39(6):469-477. doi: 10.1097/INF.0000000000002700. PMID 32398569
- [Background] Bi Q, Wu Y, Mei S, Ye C, Zou X, Zhang Z, Liu X, Wei L, Truelove SA, Zhang T, Gao W, Cheng C, Tang X, Wu X, Wu Y, Sun B, Huang S, Sun Y, Zhang J, Ma T, Lessler J, Feng T. Epidemiology and transmission of COVID-19 in 391 cases and 1286 of their close contacts in Shenzhen, China: a retrospective cohort study. Lancet Infect Dis. 2020 Aug;20(8):911-919. doi: 10.1016/S1473-3099(20)30287-5. Epub 2020 Apr 27. PMID 32353347
- [Background] Macartney K, Quinn HE, Pillsbury AJ, Koirala A, Deng L, Winkler N, Katelaris AL, O'Sullivan MVN, Dalton C, Wood N; NSW COVID-19 Schools Study Team. Transmission of SARS-CoV-2 in Australian educational settings: a prospective cohort study. Lancet Child Adolesc Health. 2020 Nov;4(11):807-816. doi: 10.1016/S2352-4642(20)30251-0. Epub 2020 Aug 3. PMID 32758454
- [Background] Perera RA, Mok CK, Tsang OT, Lv H, Ko RL, Wu NC, Yuan M, Leung WS, Chan JM, Chik TS, Choi CY, Leung K, Chan KH, Chan KC, Li KC, Wu JT, Wilson IA, Monto AS, Poon LL, Peiris M. Serological assays for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), March 2020. Euro Surveill. 2020 Apr;25(16):2000421. doi: 10.2807/1560-7917.ES.2020.25.16.2000421. PMID 32347204
- [Background] To KK, Tsang OT, Yip CC, Chan KH, Wu TC, Chan JM, Leung WS, Chik TS, Choi CY, Kandamby DH, Lung DC, Tam AR, Poon RW, Fung AY, Hung IF, Cheng VC, Chan JF, Yuen KY. Consistent Detection of 2019 Novel Coronavirus in Saliva. Clin Infect Dis. 2020 Jul 28;71(15):841-843. doi: 10.1093/cid/ciaa149. PMID 32047895
- [Background] Azzi L, Carcano G, Gianfagna F, Grossi P, Gasperina DD, Genoni A, Fasano M, Sessa F, Tettamanti L, Carinci F, Maurino V, Rossi A, Tagliabue A, Baj A. Saliva is a reliable tool to detect SARS-CoV-2. J Infect. 2020 Jul;81(1):e45-e50. doi: 10.1016/j.jinf.2020.04.005. Epub 2020 Apr 14. PMID 32298676
- [Background] Hettegger P, Huber J, Passecker K, Soldo R, Kegler U, Nohammer C, Weinhausel A. High similarity of IgG antibody profiles in blood and saliva opens opportunities for saliva based serology. PLoS One. 2019 Jun 20;14(6):e0218456. doi: 10.1371/journal.pone.0218456. eCollection 2019. PMID 31220138
- [Derived] Pinilla YT, Friessinger E, Griesbaum JM, Berner L, Heinzel C, Elsner K, Fendel R, Held J, Kreidenweiss A. Prevalence of SARS-CoV-2 Infection in Children by Antibody Detection in Saliva: Protocol for a Prospective Longitudinal Study (Coro-Buddy). JMIR Res Protoc. 2021 Oct 8;10(10):e27739. doi: 10.2196/27739. PMID 34533472